CLINICAL TRIAL: NCT00389337
Title: Sepsis: Prognosis and Evaluation of Early Diagnosis and Intervention (SPEEDI Study)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hvidovre University Hospital (Other)
Other Study IDs: KF01-108/04
Record Dates: First submitted 2006-10-17; First posted 2006-10-18 (Estimated); Last update posted 2006-10-18 (Estimated); Status verified 2006-10

CONDITIONS: SIRS; Sepsis
Keywords: Sepsis; SIRS; Biomarkers; xMAP
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
BACKGROUND: In November 2003 the Medical Director at Copenhagen University Hospital, Hvidovre, gathered a group of doctors involved in the diagnosis and treatment of patients with sepsis.

AMIS: To develop a fast and reliable tool that can guide the physician in the diagnosis and treatment of the septic patient thereby reducing mortality and morbidity. The measurement of markers of inflammation, coagulation, infection and specific bacterial antigens in the same plasma sample will give insight to the pathogenesis of sepsis and SIRS and the bodies responds to the disease.

MATERIAL AND METHODES: Case-Control study nested in cohort. 300 patients admitted to the hospital from 1.01.05 to 01.07.06. Copenhagen University Hospital, Hvidovre, an 800 beds hospital, covers a part of Copenhagen with a wide variety in the population's socioeconomic and cultural background. For the analysis of markers the luminex 100 lab analysis system is used. It utilizes xMAP® technology which enables you to simultaneously assay up to 100 analytes in a single well of a microtiter plate, using very small sample volumes. Assay development of a 15-plex is don In-house.

COWORKERS & FOUNDING: The following departments at the hospital, are coworkers in the SPEEDI study: Clinical Research Unit, Departments of Infectious Disease, Clinical Microbiology, Clinical Biochemistry, Gastroenterology (incl. surgery), Intensive Care Unit, Emergency Room, and the Hospital Board of Directors. All departments have research experience and a long tradition of publication of scientific works. The study received founding for equipment and salaries during the first phase of the study from the hospitals Board of Directors. Applications to major public foundations in Denmark are awaiting answer. No commercial interest are involved in the study.

FUTURE APPLICATIONS: A second phase of the study including children admitted at the hospital is in preparation. The very small sample volume is a great advantage in diagnosing infection in children. The applications of the study results will hopefully provide the physician with the needed tool for a fast and reliable diagnosis, prognosis and treatment guide for the patients suffering from SIRS and sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted with ≧ 2 of the following 4 symptoms of SIRS:

  * Resp. rate > 20/min
  * Heart rate > 90/min
  * Temperature > 38ºC or <36ºC
  * Leukocytes >12.000 or <4.000

Exclusion Criteria:

* Admitted to a hopital >24 h prior to inclusion
* Antibiotic therapy initiated at a hospital >8 h prior to inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2005-01; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Kofoed, MD, Principal Investigator — Copenhagen Unversity Hospital Hvidovre
Locations (1):
- Copenhagen University Hospital Hvidovre, Hvidovre, Copenhagen, Denmark

REFERENCES:
- [Derived] Kofoed K, Andersen O, Kronborg G, Tvede M, Petersen J, Eugen-Olsen J, Larsen K. Use of plasma C-reactive protein, procalcitonin, neutrophils, macrophage migration inhibitory factor, soluble urokinase-type plasminogen activator receptor, and soluble triggering receptor expressed on myeloid cells-1 in combination to diagnose infections: a prospective study. Crit Care. 2007;11(2):R38. doi: 10.1186/cc5723. PMID 17362525